CLINICAL TRIAL: NCT04376892
Title: The Effect of Exercise Capacity on Quality of Life in COPD Patients
Brief Title: Quality of Life and Exercise Capacity in COPD
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof., Izmir Katip Celebi University
Other Study IDs: IKCU2
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Copd; Quality of Life; Exercise Capacity
Keywords: copd; quality of life; exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Exercise capacity under 149 meter
  Interventions: Other: Quality of life measurement
- Group 2: Exercise capacity between 150 and 249 meter
  Interventions: Other: Quality of life measurement
- Group 3: Exercise capacity between 250 and 349 meter
  Interventions: Other: Quality of life measurement
- Group 4: Exercise capacity above 340
  Interventions: Other: Quality of life measurement

INTERVENTIONS:
Other: Quality of life measurement — Quality of life measurement by St. George Respiratory questionnaire

SUMMARY:
COPD patients will be examined in 4 groups according to their walking distance. Patients walking under 150 meters will be determined as Group 1, those walking between 150-249 meters will be Group 2, those walking between 250-349 meters will be selected as Group 3, and patients with COPD who walk 350 and above will be determined as Group 4. The groups were compared in terms of quality of life, psychological symptoms and dyspnea.

DETAILED DESCRIPTION:
Quality of life affects the mortality rate independently in patients with COPD. The treatment applied in COPD does not stop the decrease in lung function, nor does it prolong the survival time. Spirometric evaluations to determine the severity of the disease are not sufficient to explain the perception of patients and their adaptation to their diseases. Therefore, evaluating the quality of life has become an important measure of treatment in COPD patients. Quality of life measurements should be done to minimize the effect of the disease, to help patients better cope with the consequences of an incurable long-term condition, and to determine modifiable factors. Identifying modifiable factors; in personalized treatment adopted in airway diseases in recent years; it is important to be able to apply appropriate pharmacological and non-pharmacological treatments Our aim is to exercise capacity in COPD patients; firstly to investigate the effect on quality of life, then to determine the relationship between emergency admission and hospitalization, dyspnea, psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients completed all tests and qustionnaires

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Above 18
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | 20 minutes
  St. George Respiratory Questionnaire

SECONDARY OUTCOMES:
Dyspnea Severity | 5 minutes
  mMRC
Respiratory Function | 20 minutes
  Respiratory Function Test
Anxiety Depression | 20 minutes
  Hospital anxiety and Depression Qustionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hulya S, Ilknur N, Gulru P. Effect of exercise capacity on perception of dyspnea, psychological symptoms and quality of life in patients with chronic obstructive pulmonary disease. Heart Lung. 2020 Nov-Dec;49(6):753-757. doi: 10.1016/j.hrtlng.2020.09.008. Epub 2020 Sep 23. PMID 32979640